CLINICAL TRIAL: NCT05883774
Title: Effects of Repetitive Transcranial Magnetic Stimulation on the Anxiety State of Older Patients With Generalized Anxiety Disorder
Brief Title: Effects of rTMS on the Anxiety State of Older Patients With GAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS-GAD
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: repetitive transcranial magnetic stimulation; generalized anxiety disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS (Active Comparator): Patients are treated with repetitive transcranial magnetic stimulation (rTMS).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- sham-rTMS (Sham Comparator): Patients are treated with sham repetitive transcranial magnetic stimulation (sham-rTMS).
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS is applied using a transcranial magnetic stimulator with a figure-of-8 coil once per day for 10 consecutive days. rTMS is delivered to the right dorsolateral prefrontal cortex (DLPFC) at a frequency of 1 Hz for 20 minutes (1200 total pulses).
  Other Names: rTMS
  Arms: rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation — Sham-rTMS is performed in the same way as the treatment group except that the coil is rotated 90° away from the scalp.
  Other Names: sham-rTMS
  Arms: sham-rTMS

SUMMARY:
The purpose of this study is to evaluate the effects of low-frequency repetitive transcranial magnetic stimulation on anxiety state in older patients with generalized anxiety disorder.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation can alter nerve cell excitability, improve cerebral blood flow and metabolism, and is widely used in neuropsychiatric research. Studies have shown its efficiency and safety in treating anxiety disorders, however the senior patient group has not been adequately validated. The purpose of this study is to evaluate the effects of low-frequency repetitive transcranial magnetic stimulation on anxiety state in older patients with generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* 1）Age≥60 years, regardless of gender.
* 2）Meets the diagnostic criteria for generalized anxiety disorder in the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) developed by the American Psychiatric Association.
* 3）HAMA score≥14 and HAMD-17 items score <17.
* 4）No adjustment in the type and dose of anti-anxiety medication in the 3 months prior to randomization.
* 5）Willing to participate and sign the informed consent.

Exclusion Criteria:

* 1）Traumatic brain injury or other conditions affecting the brain, such encephalitis, brain tumors, or intracranial hypertension.
* 2）Previous history of epilepsy, family history of epilepsy or presence of seizure provoking factors or alcohol abuse.
* 3）History of other psychiatric disorders such as current post-traumatic stress disorder, substance use disorder (within 6 months), bipolar disorder and obsessive-compulsive disorder.
* 4）Unstable mental state with impulses toward self-harm or suicide.
* 5）Presence of intracranial metal implant, cochlear implant, built-in pulse generator (such as cardiac pacemaker), etc.
* 6）Medical or surgical disorders that are severe or unstable.
* 7）Pregnancy or breastfeeding.
* 8) Those who are participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to enrollment.
* 9) Other conditions that the researchers think are not suitable for the project.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Differences in HAMA scores after 10 sessions of rTMS/sham-rTMS between two groups. | baseline; 10 days
  The HAMA scale consists of 14 items, each with a score ranging from 1 to 4, for a total score ranging from 14 to 56, and the degree of anxiety correlates positively with the score.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China